CLINICAL TRIAL: NCT04346732
Title: Effectiveness of Vapocoolant Spray on Venipuncture Pain in Young Male Donors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Semra Aciksoz, Assistant Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SAciksoz
Record Dates: First submitted 2020-04-11; First posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Venipuncture; Pain
Keywords: Vapocoolant Spray; Venipuncture; Pain; Donors
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The participants were separated into two groups with the randomisation method.These groups were named the vapocoolant spray group and the control group
Who Masked: Investigator
Masking Description: In both groups, immediately following venipuncture, pain assessment was made with the VAS by the researcher, who did not know which group each participant belonged to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vapocoolant spray (Experimental): Vapocoolant spray was applied to the donors in the vapocoolant spray group.
  Interventions: Other: Vapocoolant spray
- Control (No Intervention): The donors in the control group were not given any intervention during the blood collection process.

INTERVENTIONS:
Other: Vapocoolant spray — Vapocoolant spray
  Arms: Vapocoolant spray

SUMMARY:
Aim: The aim of this study is to assess the effectiveness of vapocoolant spray in reducing pain related to venipuncture in young, healthy male blood donors.

Hypotheses:

H1: Vapocoolant spray reduces venipuncture pain during blood donation. H0: Vapocoolant spray does not reduce venipuncture pain during blood donation.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent. Before the procedure was begun, the donors who agreed to participate in the study were met face-to-face and asked to fill in the "Informative Characteristics Form", the "VAS", the "Blood/Injection Fear Scale" and the "STAI-I" forms.Then the donors were assigned to their groups by the researcher.The donors in the control group were not given any intervention during the blood collection process. Vapocoolant spray was applied to the donors in the vapocoolant spray group. During the blood collection procedure, after the donors' skin was cleaned with antiseptic solution, spray was applied to the application site for a maximum of 10-15 seconds from a distance of 25 cm. In both groups, immediately following venipuncture, pain assessment was made with the VAS by the researcher, who did not know which group each participant belonged to.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 35
* BMI between 18.5 and 24.9 kg/m2
* speaks turkish
* male donor
* individuals who applied to make voluntary blood donations
* volunteers to participate in the study

Exclusion Criteria:

* donors who did not agree to take part in the study,
* donors with open wound, scar, infection, dermatitis, eczema or lesion at the venipuncture site, or donors with cold allergy

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in venipuncture pain on the Visual Analogue Scale(VAS) during blood donation | immediately following venipuncture procedure
  The VAS is used to inquire about pain levels resulting from venipuncture.In the 10 cm-long VAS, 0 indicates no pain, while 10 indicates the most intense pain.